CLINICAL TRIAL: NCT04346264
Title: CoVid-19 - Infection and Antibody Formation in the Viennese Population - Data From the Vienna Health Study LEAD
Brief Title: CoVid-19 - Infection and Antibody Formation in the Viennese Population
Status: Completed | Type: Observational
Sponsor: Ludwig Boltzmann Institute for Lung Health (Other)
Responsible Party: Sponsor
Other Study IDs: LEAD CoVid-19
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Virus Diseases; COVID-19
MeSH Terms: conditions — Virus Diseases; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- General Cohort: Population general cohort from the Austrian LEAD Study
  Interventions: Diagnostic Test: NO intervention planned due to the observational study design only a diagnostic testing

INTERVENTIONS:
Diagnostic Test: NO intervention planned due to the observational study design only a diagnostic testing — Only a diagnostic test (serum blood and antibody measurement) is planned

SUMMARY:
Summary of the study

Study population:

A representative sample of the Viennese population stratified by age and gender (data from the Vienna Health Study LEAD)

Potential output and analysis:

* Extent of age-specific infection and antibody formation
* Cumulative incidence of infection
* Rate of asymptomatic infection
* Relationship with socioeconomics, lifestyle and risk factors (comorbidities)

Study design:

Prospective, longitudinal, stratified by age and gender

Duration of study:

Initial testing as soon as possible and repeat based on monitoring of the pandemic curve (probably after 2-3 months)

Information to be obtained from participants:

* serum samples for information on SARS-CoV2 infection and antibody formation
* data on clinical symptoms

DETAILED DESCRIPTION:
Both international (WHO; (1) and national are calling for increased testing for the SARS-CoV-2 virus; at present it is completely unclear how many people will actually become infected with the Covid-19 virus or have formed antibodies against it during the pandemic. The greatest uncertainty of all calculation models on hospitalisation rates, morbidity and mortality of the pandemic is the unknown number of unreported cases of citizens infected or having been infected with Covid-19.

Currently the direct detection of the SARS-CoV-2 virus from the mouth/nose/throat swab using PCR is established worldwide with high sensitivity and specificity. This direct method is expensive and not always available in sufficient quantities. Furthermore, the results are strongly influenced by the quality of the smear collection.

The detection of antibodies against the SARS-CoV-2 virus is an alternative method for determining whether a person has been infected with SARS-CoV-2 and has developed an immune response to the virus. Recently several companies have been offering such kits for sale. According to national experts, these kits have not yet been sufficiently clinically validated, which is why valid data on their sensitivity and specificity are not yet available. However, on the validation of these tests are being worked hard all over the world, so that it can be assumed (the experts also agree on this) that data on the sensitivity and specificity of the antibody tests will be available in the foreseeable future.

Probably the only reasonable and feasible method of testing the actual rate of Covid-19 infection in a given population is to detect infection (either directly or indirectly by means of antibody testing) from a sample that is as representative as possible for this population.

The selected subjects of the LEAD study, the core project of the Ludwig Boltzmann Institute for Lung Health at Otto Wagner Hospital (the hospital association is an official partner of the institute), represent an exemplary representative sample of the general population in Vienna (i.e. the sample corresponds to the Viennese population in terms of age, gender, smoking habits, place of residence, etc.). In the LEAD study, more than 11,000 subjects (aged 6-80) mainly from Vienna were subjected to a "Health examination survey" (2).

Due to the conditions described above, blood should be drawn from the subjects of the LEAD study at two points in time (as early as possible and after two to three months) and blood sera should be frozen to determine antibodies against SARS-CoV-2 and tested with a test of high sensitivity and specificity. According to the WHO this procedure (longitudinal cohort study with serial sampling of the same individuals (in the same geographic area) each time) is recommended in that provides the most comprehensive information on extent of infection.

By testing for SARS-CoV-2 antibodies twice in the subjects of the LEAD study (random sample), an accurate and representative estimate of the actual positive Covid-19 cases in the Viennese population and the rate of spread during the pandemic could be extrapolated for Vienna in the foreseeable future. Since more than 1,500 individual parameters were measured in the participants of the LEAD study, conclusions on socioeconomics, lifestyle factors and possible risk profiles (e.g. co-morbidity, smoking behaviour, etc.) can be drawn from those who tested positive (but also negative). In addition, a query regarding symptoms should be carried out at both dates in order to obtain information on the percentage of asymptomatic infections with SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria: all participants of the Austrian LEAD study will be invited (www.leadstudy.at) -

Exclusion Criteria: pregnancy, failure due to language

-

Ages: 6 Years to 85 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: General population cohort (The Austrian LEAD Study, NCT01727518), aged 6-85 years from Vienna, Austria
Sampling Method: Probability Sample
Enrollment: 12419 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 antibody titres | 5 weeks
  Antibody Titres IgG and IgM

SECONDARY OUTCOMES:
Prevalence of SARS-CoV-2 antibody titres after 3 Months | 4 Months
  Re-Calculation including incidence of the general population

CONTACTS AND LOCATIONS:
Overall Officials: Otto C Burghuber, Prof.MD, Principal Investigator — Ludwig Boltzmann Institute for Lung Health
Locations (1):
- The LEAD Study Center, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Breyer-Kohansal R, Faner R, Breyer MK, Ofenheimer A, Schrott A, Studnicka M, Wouters EFM, Burghuber OC, Hartl S, Agusti A. Factors Associated with Low Lung Function in Different Age Bins in the General Population. Am J Respir Crit Care Med. 2020 Jul 15;202(2):292-296. doi: 10.1164/rccm.202001-0172LE. No abstract available. PMID 32255673
- See also: Homepage of the Austrian LEAD Study — http://www.leadstudy.at